CLINICAL TRIAL: NCT05820880
Title: Evaluation of the Clinical Efficacy and Safety of Perindopril 5 mg / Indapamide 1.25 mg / Amlodipine 5 mg Fixed Combination in Single-pill After 2 Months of Treatment Versus Free Combination, Perindopril 4 mg / Indapamide 1.25 mg + Amlodipine 5 mg Given Separately at the Same Time, With Conditional Titration Based on Blood Pressure Control in Patients With Essential Hypertension Uncontrolled After 1 Month With Perindopril 4 mg / Indapamide 1.25 mg Bi-therapy.
Brief Title: Efficacy and Safety of Perindopril 5 mg / Indapamide 1.25 mg / Amlodipine 5 mg Fixed Combination in Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL3-6593-018
Record Dates: First submitted 2023-02-28; First posted 2023-04-20 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fixed [Per/Ind/Aml] (Experimental): From inclusion to Month 2, patients receive the fixed combination of perindopril 5 mg / indapamide 1.25 mg / amlodipine 5 mg (S06593).
  From Month 2 to 4, patients either stay at the same dose if the blood pressure is controlled, either are up-titrated to the next dose of the strategy if the blood pressure is not controlled (ie, perindopril 10 mg / indapamide 2.5 mg / amlodipine 5 mg).
  From Month 4 to 6, patients either stay at the same dose if the blood pressure is controlled, either are up-titrated to the next dose of the strategy if the blood pressure is not controlled (ie, for patients who were up-titrated at Month 2 visit: perindopril 10 mg / indapamide 2.5 mg / amlodipine 10 mg or for patients who were not yet up-titrated: perindopril 10 mg / indapamide 2.5 mg / amlodipine 5 mg.
  Interventions: Drug: Fixed [Per/Ind/Aml]
- Free [Per/Ind + Aml] (Active Comparator): From inclusion to Month 2, patients receive the free combination of perindopril 4 mg / indapamide 1.25 mg plus amlodipine 5 mg.
  From Month 2 to 4, patients either stay at the same dose if the blood pressure is controlled, either are up-titrated to the next dose of the strategy if the blood pressure is not controlled (ie, double dose of perindopril 4 mg / indapamide 1.25 mg plus amlodipine 5 mg for patients).
  From Month 4 to 6, patients either stay at the same dose if the blood pressure is controlled, either are up-titrated to the next dose of the strategy if the blood pressure is not controlled (ie for patients who were up-titrated at Month 2 visit: double dose of perindopril 4 mg / indapamide 1.25 mg plus double dose of amlodipine 5 mg or for patients who were not yet up-titrated:double dose of perindopril 4 mg / indapamide 1.25 mg plus amlodipine 5 mg.
  Interventions: Drug: Free [Per/Ind + Aml]

INTERVENTIONS:
Drug: Fixed [Per/Ind/Aml] — Fixed Dose combination of Perindopril/Indapamide/Amlodipine
  Arms: Fixed [Per/Ind/Aml]
Drug: Free [Per/Ind + Aml] — Free dose combination of Perindopril/Indapamide and Amlodipine
  Arms: Free [Per/Ind + Aml]

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of a fixed-dose combination of perindopril 5 mg /indapamide 1.25 mg / amlodipine 5 mg compared to the free combination of the same components (perindopril 4 mg / indapamide 1.25 mg in a single pill and amlodipine 5 mg pill given separately at the same time) in chinese patients with uncontrolled essential hypertension.

ELIGIBILITY:
Main Inclusion Criteria:

* Men or women of Asian origin
* ≥18 years old
* Treated for essential hypertension
* Having the day of the selection visit an uncontrolled hypertension treated with any anti-hypertensive monotherapy at maximal dose or any dual therapy at starting dose according to investigator's routine practice or at least 1 month prior to the visit
* Having at the selection visit a sitting SBP≥140 and <180 mmHg and DBP≥90 and <110 mmHg

Main Exclusion Criteria:

* Known or suspected symptomatic orthostatic hypotension or positive orthostatic test at the selection visit
* Treatment with more than 2 antihypertensive drugs or with 2 antihypertensive drugs at the highest doses at the selection visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 532 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2022-02-23 (Actual)

PRIMARY OUTCOMES:
Sitting SBP change after two months of treatment | Baseline safety visit, Month 2 follow-up visit
  Office sitting Systolic Blood Pressure (SBP) change from baseline to last post-baseline value over the period from Month 0 to month 2

SECONDARY OUTCOMES:
Sitting SBP change from month 2 to month 4 | Month 2 follow-up visit, Month 4 follow-up visit
  Office sitting Systolic Blood Pressure (SBP) change from month 2 to month 4
Sitting SBP change from month 4 to month 6 | Month 4 follow-up visit, Month 6 follow-up visit
  Office sitting Systolic Blood Pressure (SBP) change from month 4 to month 6
Sitting DBP change after two months of treatment | Baseline safety visit, Month 2 follow-up visit
  Office sitting Diastolic Blood Pressure (DBP) change from baseline to last post-baseline value over the period from Month 0 to month 2
Sitting DBP change from month 2 to month 4 | Month 2 follow-up visit, Month 4 follow-up visit
  Office sitting Diastolic Blood Pressure (DBP) change from month 2 to month 4
Sitting DBP change from month 4 to month 6 | Month 4 follow-up visit, Month 6 follow-up visit
  Office sitting Diastolic Blood Pressure (DBP) change from month 4 to month 6
Sitting Mean Arterial Pressure change after two months of treatment | Baseline safety visit, Month 2 follow-up visit
  Sitting Mean Arterial Pressure (MAP) change from baseline to last post-baseline value over the period from Month 0 to month 2 with MAP=2/3 DBP+1/3 SBP
Sitting Mean Arterial Pressure change from month 2 to month 4 | Month 2 follow-up visit, Month 4 follow-up visit
  Sitting Mean Arterial Pressure (MAP) change from from month 2 to month 4 , with MAP=2/3 DBP+1/3 SBP
Sitting Mean Arterial Pressure change from month 4 to month 6 | Month 4 follow-up visit, Month 6 follow-up visit
  Sitting Mean Arterial Pressure (MAP) change from from month 4 to month 6, with MAP=2/3 DBP+1/3 SBP
Sitting Pulse Pressure change after two months of treatment | Baseline safety visit, Month 2 follow-up visit
  Sitting Pulse Pressure change from baseline to last post-baseline value over the period from Month 0 to month 2, with Pulse Pressure=SBP-DBP
Response to the treatment at two months | Month 2 follow-up visit
  Number of patients responders, ie: with control of Blood Pressure : sitting SBP <140 mmHg and sitting DBP <90 mmHg) and/or sitting SBP decrease from baseline ≥20 mmHg or sitting DBP decrease from baseline ≥10 mmHg.
Control of Blood Pressure at two months | Month 2 follow-up visit
  Number of patients with Blood pressure controlled, ie : with sitting SBP <140 mmHg and sitting DBP < 90 mmHg
Adverse events between Month 0 and Month 2 | Up to the 2 month follow-up visit
  Number experiencing treatment emergent adverse events between month 0 and month 2
Adverse events between Month 0 and Month 6 | Up to the 6 month final visit
  Number experiencing treatment emergent adverse events between month 0 and month 6

CONTACTS AND LOCATIONS:
Locations (42):
- China (42):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Xuanwu Hospital Capital Medical Universtiy, Beijing, Beijing Municipality
  - The First affiliated hospital Chongqing Medical University, Chongqing, Chongqing Municipality
  - The second affiliated hospital of Chongqing medical university, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The first affiliated hospital of Fujian medical university, Fuzhou, Fujian
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First affiliated hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First affiliated hospital of Zhengzhou University, Zhengzhou, Henan
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hosptial of Baotou Medical college, Innter Mongolia University of Science & Technology, Baotou, Inner Mongolia
  - Inner Mongolia People's Hospital, Hohhot, Inner Mongolia
  - The Affiliated Hospital of Xuzhou Medical College, Xuzhou, Jiangshu
  - Xuzhou Central Hospital, Xuzhou, Jiangshu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Wuxi Second People's Hospital, Wuxi, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - Yangzhou First People's Hospital, Yangzhou, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - The First affiliated hospital of Nanchang University, Nanchang, Jiangxi
  - The Second affiliated hospital of Nanchang University, Nanchang, Jiangxi
  - Jilin university China-Japan Union Hospital, Changchun, Jilin
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - Daqing Oilfield general hospital, Daqing, Liaonig
  - First affiliated hospital of Dalian medical university, Dalian, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - The People's Hospital of Liaoning Province, Shenyang, Liaoning
  - The Affiliated Jiangning Hospital of Nanjing Medical University, Nanjing, Nanjing
  - Qinghai Provincial People's Hospital, Xining, Qinghai
  - Shandong Provincial Qianfoshan Hospita, Jinan, Shandong
  - Linyi People's Hospital, Linyi, Shandong
  - Zaozhuang Municipal Hospital, Zaozhuang, Shandong
  - Ruijin Hospital affiliated to Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - The First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The First Affiliated Hospital, School of Medicine of Xi'an Jiaotong University, Xi’an, Shanxi
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Tianjin People's hospital, Tianjin, Tianjin Municipality
  - People's Hospital of Xinjiang Uyghur Autonomous Region, Ürümqi, Uyghur Autonomous Region

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1st January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: https://clinicaltrials.servier.com/

REFERENCES:
- [Background] Wang JG, Topouchian J, Bricout-Hennel S, Mu J, Chen L, Li P, He S, Luo S, Jiang W, Jiang Y, Sun Y, Zhang Y, Asmar R. Efficacy and safety of a single-pill versus free combination of perindopril/indapamide/amlodipine: a multicenter, randomized, double-blind study in Chinese patients with hypertension. J Hypertens. 2024 Aug 1;42(8):1373-1381. doi: 10.1097/HJH.0000000000003741. Epub 2024 Apr 24. PMID 38660708